CLINICAL TRIAL: NCT03545880
Title: Effects of Kinesiotaping on Post-Needling Soreness by Dry Needling on Active Trigger Points
Brief Title: Kinesiotaping and Post-dry Needling Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Director of Department, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URJC 2018-12
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Mechanical Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping (Experimental): A Kinesiotaping will be provided over the upper trapezius muscle after the application of dry needling
  Interventions: Other: Kinesiotaping
- Placebo (Placebo Comparator): Individuals will not perform any action after the application of trigger point dry needling
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Kinesiotaping — A Kinesiotaping will be provided over the upper trapezius muscle after the application of dry needling
  Arms: Kinesiotaping
Other: Placebo — Individuals will not perform any action after the application of trigger point dry needling
  Arms: Placebo

SUMMARY:
Application of trigger point dry needling can induce post-dry needling soreness. This is not a negative experience, but sometimes some patients want to reduce it as much as possible. Different therapeutic strategies targeting to decrease post-dry needling soreness need to be investigated. Since Kinesiotaping has been advocated for decreasing tone in the muscle tissues, it would be a potential intervention for this objective.

ELIGIBILITY:
Inclusion Criteria:

- Generalized neck-shoulder pain with symptoms provoked by neck postures, neck movement, or palpation of the cervical musculature

Exclusion Criteria:

* any contraindication to dry needling
* whiplash injury;
* previous cervical surgery;
* cervical radiculopathy or myelopathy;
* diagnosis of fibromyalgia syndrome;
* having undergone any therapy intervention for the neck are in the previous 6 months;
* fear to needles;
* less than 18 or greater than 65 years of age.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-08-05 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Changes in post-dry needling pain intensity before and after the intervention | Baseline, immediately after, 24 hours after, 48 hours after and 72 hours after treatment
  A Numerical Pain Rate Scale (NPRS, 0-10) will be used to record post-dry needling soreness and pain

SECONDARY OUTCOMES:
Changes in cervical related-disability before and after the intervention | Baseline and 72 hours after treatment
  The Neck Disability Index (NDI) will be used
Changes in upper extremity related-disability before and after the intervention | Baseline and 72 hours after treatment
  The Shoulder Pain and Disability Index (SPADI) questionnaire will be used
Changes in pressure pain sensitivity | Baseline, immediately after and 72 hours after treatment
  Pressure pain threshold over the Trigger Point area will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain